CLINICAL TRIAL: NCT00908440
Title: Decision Aid in Veterans With Posttraumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Bradley Vince Watts, MD, MPH, White River Junction VAMC
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 07-266
Record Dates: First submitted 2009-05-20; First posted 2009-05-25 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Decision Aid; Posttraumatic Stress Disorder; evidence-based treatments
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Decision Aid — 25 page booklet informing patients about PTSD symptoms and treatment options

SUMMARY:
The purpose of this study is to examine the effects of a decision aid on veterans with posttraumatic stress disorder (PTSD) presenting for care. The investigators' primary hypothesis is that patients assigned to use the decision aid will demonstrate improved quality of decisions regarding PTSD treatment relative to patients assigned to usual care. Improved decision quality will be examined by assessing patient's knowledge of treatments, evaluation of the risk and benefits, ability to arrive at a decision, and certainty about that decision. The investigators' secondary hypothesis is that patients assigned to the decision aid will be more satisfied with their care and more compliant with their care compared to patients assigned to receive usual care. The investigators will also determine whether patients assigned to the decision aid, relative to patients assigned to usual care, are more likely to receive evidence-based treatments for PTSD and experience reductions in PTSD symptoms.

DETAILED DESCRIPTION:
Posttraumatic stress is a severe and often disabling condition affecting millions of veterans. Within VA, significant staffing and financial resources are devoted to the mission of treating PTSD and the anticipated need for treatment is expected to accelerate as veterans return from the Iraq war.

Research has identified a number of successful strategies for the treatment of PTSD, including both psychotherapy and pharmacology. Several treatments, including group psychotherapy and benzodiazepines have demonstrated a lack of efficacy in the treatment of PTSD. Despite this knowledge, many veterans with PTSD do not receive an evidence-based treatment and may even receive a treatment known to not be effective. Among the group of proven effective treatments, the patient time commitment and adverse effects differ considerably. Patients with PTSD are often ill informed about the available treatments, and there has been little formal effort aimed at matching the patients' preferences to a specific treatment.

We propose to conduct a clinical trial of a decision aid for veterans with PTSD. Decision aids are standardized, evidence-based tools to help patients choose between two or more preference-sensitive, clinically acceptable options when there is no clear "best" option. Decision aids are designed to provide patients with detailed balanced information about all the viable treatment options. In addition, they seek to assist the patient in clarifying their own values and preferences such that the patient may choose among the available treatment options.

We believe that the use of a decision aid, compared to treatment as usual, will result in a more patient-centered approach that ultimately will increase the likelihood of the patient receiving evidence based care, both of which are priority goals of VHA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who meet criteria for Posttraumatic Stress Disorder on the Posttraumatic Stress Disorder Checklist (PCL).

Exclusion Criteria:

* Patients must not have active substance abuse.
* Patients must not have received VA PTSD treatment within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge of treatments, evaluation of the risk and benefits, as assessed by the Knowledge Questionnaire | 1 week
Ability to arrive at a decision and certainty about that decision, score on the Decisional Conflict Scale | 1 week
Satisfaction with care and compliance with care, score on the Survey of Health Experiences | 1 week

SECONDARY OUTCOMES:
Use of evidence based treatments and overall cost | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bradley V Watts, MD, MPH, Principal Investigator — White River Junction Veterans Affairs Medical Center; Paula Schnurr, PHD, Principal Investigator — White River Junction Veterans Affairs Medical Center
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States

REFERENCES:
- [Background] Foa, E.B., Keane, TM, Friedman, M.J. (eds): Effective treatments for PTSD: Practice guidelines from the International Society for Traumatic Stress Studies. NY, Guilford, 2000.
- [Background] Watts, B., Mayo, L., Weeks, W. A meta analysis of treatments for posttraumatic stress disorder, in International Society for Traumatic Stress Studies 21st Annual meeting. Toronto, Canada, 2005.
- [Background] O'Connor AM, Stacey D, Entwistle V, Llewellyn-Thomas H, Rovner D, Holmes-Rovner M, Tait V, Tetroe J, Fiset V, Barry M, Jones J. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2003;(2):CD001431. doi: 10.1002/14651858.CD001431. PMID 12804407
- [Background] Rosen CS, Chow HC, Finney JF, Greenbaum MA, Moos RH, Sheikh JI, Yesavage JA. VA practice patterns and practice guidelines for treating posttraumatic stress disorder. J Trauma Stress. 2004 Jun;17(3):213-22. doi: 10.1023/B:JOTS.0000029264.23878.53. PMID 15253093
- [Derived] Watts BV, Zayed MH, Llewellyn-Thomas H, Schnurr PP. Understanding and meeting information needs for patients with posttraumatic stress disorder. BMC Psychiatry. 2016 Feb 1;16:21. doi: 10.1186/s12888-016-0724-x. PMID 26830930